CLINICAL TRIAL: NCT06290557
Title: A Randomized Double-blind Placebo-controlled First-in-man Single-dose and Multiple Dose Study to Evaluate the Safety, Tolerability and Efficacy of a Recombinant Chimeric Bacteriophage Endolysin HY-133 With an Extended Phase to Evaluate Effects of the Nasal Microbiome
Brief Title: First-in-man Single-dose and Multiple Dose Study to Evaluate the Safety, Tolerability and Efficacy ofHY-133
Acronym: HY-133
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HY-133; 2023-507737-17-00 (EU CTIS Number)
Record Dates: First submitted 2024-02-22; First posted 2024-03-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Staphylococcus Aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Low Dose single application Low Dose multiple application High Dose single application high dose multiple application
  Interventions: Drug: HY_133
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HY_133 — A recombinant chimeric bacteriophage endolysin HY-133
  Arms: Verum
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In this clinical trial we will test a new approach for decolonization of S. aureus.

As innovative product HY-133 a recombinant chimeric bacteriophage endolysin will be sprayed in both nostrils of healthy subjects once or five times in one day. To avoid possible bias the subjects will be randomized 3:2 verum vs placebo, moreover the subject as well as the investigator will be blinded to the group assigned.

ELIGIBILITY:
Inclusion Criteria

* Must be ≥ 18 years at the time of signing the informedconsent.
* Understand and voluntarily sign an informed consent document prior to any study related
* assessments/procedures.
* Nasal colonization with methicillin-susceptible S. aureus (MSSA)
* Female Subject of childbearing potential1 and male subjects with female partner of childbearing potential1 is willing to use highly effective contraceptive methods during treatment until end of study at D15

Exclusion Criteria

* Nasal colonization with methicillin-resistant S. aureus (MRSA)
* Nasal traumata including nose penetrating foreign bodies (e.g. piercings)
* Presence of any significant morbidity, e.g. Diabetes, cardiovascular disease
* Acute or known chronic diseases of the nose or the paranasal sinuses
* Acute or known chronic diseases of other parts of the respiratory tract
* Running nose due to other reasons (e.g. allergic diseases)7. Positive serological HIV, hepatitis A, B or C test. In case of positive HBsAg, volunteer must provide prove of hepatitis B vaccination, otherwise volunteer must be excluded.
* Women during pregnancy and lactation.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* Participation in other clinical trials or observation period of competing trials, in the 12 weeks prior to screening.
* Acute or chronic, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the Investigator based on medical history, physical exam, and/or laboratory screening test
* Systemic antibiotic treatment in the 12 weeks prior to screening.
* Intranasal eradication therapy in the 12 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
ADRs/AEs/SAEs occurring from the time of application until the final study visit (Day15) for each subject | baseline, pre-intervention/procedure/surgery, up to Day15
  The primary objective of this trial is to evaluate the safety of the HY-133. Fort the primary objective the nature, frequency, and severity of AEs and/or SAEs occurring in the study are recorded as follows: ADRs/AEs/SAEs occurring from the time of application until the final study visit (D15) for each subject A DLT is defined as any AE of Grade 4 or above related to the IMP

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Department of Dermatology, University Hospital Tuebingen, Tübingen
  - Department of Dermatology, Tübingen